CLINICAL TRIAL: NCT05452486
Title: Comparing Central Auditory Processing Performance in Bilinguals Using L1 vs. L2 Materials
Brief Title: Auditory Processing in Spanish-English Bilinguals: Is Performance Better When Tested in Spanish or English?
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: University of Arkansas (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Crossover | Masking: None | Purpose: Diagnostic
Other Study IDs: 274429
Record Dates: First submitted 2022-07-06; First posted 2022-07-11 (Actual); Results first posted 2024-09-19 (Actual); Last update posted 2024-09-19 (Actual); Status verified 2024-05

CONDITIONS: Auditory Processing Disorder
Keywords: bilingual; Spanish
MeSH Terms: conditions — Auditory Perceptual Disorders

STUDY DESIGN:
Intervention Model Description: This study is a repeated measures experimental design in which participants will complete auditory processing tests in both English (L2) and Spanish (L1). The presentation of Spanish and English test materials will be counterbalanced across participants to minimize fatigue and practice effects.
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- L1 First (Experimental): All participants will receive both experimental conditions (i.e., test materials in English, test materials in Spanish) in a counterbalanced order. Individuals in this arm receive Spanish materials first, then English test materials.
  Interventions: Diagnostic Test: English APD assessment; Diagnostic Test: Spanish APD assessment
- L2 First (Experimental): All participants will receive both experimental conditions (i.e., test materials in English, test materials in Spanish) in a counterbalanced order. Individuals in this arm receive English materials first, then Spanish test materials.
  Interventions: Diagnostic Test: English APD assessment; Diagnostic Test: Spanish APD assessment

INTERVENTIONS:
Diagnostic Test: English APD assessment — Materials presented in English
Diagnostic Test: Spanish APD assessment — Materials presented in Spanish

SUMMARY:
The purpose of this study is to learn more about how bilingual individuals process sound in challenging listening environments and how testing language may impact results on auditory processing assessments. Auditory processing evaluations assess specific auditory skills necessary to hear and understand complex auditory signals, but many of these tests rely heavily on language. This poses an issue for individuals with native languages other than English because the test results may not clearly identify whether performance is due to an auditory processing problem or to the language used in the test materials. This study aims to identify whether auditory processing performance differs in Spanish-English bilinguals based on the language of the test materials used (English vs. Spanish). Ultimately, the results of this study may aid in more accurate diagnoses and treatment of auditory processing disorders in bilingual individuals.

DETAILED DESCRIPTION:
Auditory processing disorder (APD) is a disorder caused by a disruption within the central auditory pathway that impairs processing of complex or degraded auditory inputs. Patients with this condition often present with normal hearing but still report problems understanding speech. This commonly manifests as individuals having difficulty understanding speech in challenging listening environments (e.g., noisy backgrounds, reverberant environments, rapid speech), localizing sounds, and following complex auditory directions. An underlying auditory skill vital to these processes is binaural processing, or the ability to utilize auditory cues from both ears. Binaural processing aids in identifying a talker in the midst of background noise and allows us to better separate relevant from irrelevant inputs.

While auditory processing evaluations assess specific auditory skills (like binaural processing) necessary for efficient processing and understanding of complex auditory signals, many of the tests rely heavily on language. This poses an issue for individuals for whom English is not their native language. Because the tests are linguistically loaded, the obtained results do not clearly identify whether an issue should be attributed to a central auditory problem or to the language used in the test materials. Thus, audiologists are often hesitant to test bilingual patients who demonstrate features of APD.

It is possible that bilingual individuals would perform more favorably when tested in their native language (L1). Indeed, differences in complex auditory task performance have been seen in Spanish-English bilinguals when materials were presented in Spanish versus English. Recent studies have evaluated test-language effects in bilingual education and described significant improvements in performance when bilinguals were instructed and tested in their native language (L1) compared to performance in their later acquired language (L2). Numerous studies have also assessed monolingual vs. bilingual performance in complex auditory tasks including listening in noise, auditory memory, and competing speech. While much research in auditory processing of bilingual speakers compares performance between monolinguals and bilinguals, evidence to inform best clinical practice in the assessment of APD in bilinguals is lacking. To date, relatively few studies investigate performance within the same participant with testing language being the differential factor.

Therefore, the purpose of this study is to compare binaural processing performance in Spanish-English bilingual participants when tested in Spanish (L1) versus in English (L2). Based on prior literature, we suspect that bilingual participants will perform better when they are instructed and presented with assessments in their native language versus when they are assessed in their later acquired language (L2). However, it is possible that our participants, who will be proficient in both L1 and L2, will show no difference in task performance. Regardless, by comparing binaural processing performance in bilingual participants, we will clarify whether testing bilingual individuals in a secondary language (when proficient in that language) results in valid and reliable measures of their auditory processing abilities. Thus, our results will provide evidence to establish best clinical practice when evaluating bilingual listeners for auditory processing deficits. This will enable clinicians to more confidently evaluate and diagnose auditory processing disorders in bilingual populations.

ELIGIBILITY:
Inclusion Criteria:

* Bilingual Spanish-English speakers
* Must have learned Spanish first followed by English
* Proficiency in both languages
* Normal hearing

Exclusion Criteria:

* Hearing loss
* History of traumatic brain injuries (TBI)
* Neurological issues
* Auditory processing concerns

Ages: 18 Years to 55 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult
Enrollment: 29 (Actual)
Dates: Start 2022-07-25 (Actual); Primary Completion 2022-11-16 (Actual); Study Completion 2022-11-16 (Actual)

CONTACTS AND LOCATIONS:
Locations (1):
- University of Arkansas for Medical Sciences, Little Rock, Arkansas, United States

IPD SHARING:
Plan to Share IPD: Undecided

REFERENCES:
- [Background] American Speech-Language-Hearing Association. (n.d.). Central Auditory Processing Disorder. (Practice Portal). Retrieved May 17, 2022, from www.asha.org/Practice-Portal/Clinical-Topics/Central-Auditory-Processing-Disorder/.
- [Background] Canz, T., Piesche, N., Dallinger, S., & Jonkmann, K. (2021). Test-language effects in bilingual education: Evidence from CLIL classes in Germany. Learning and Instruction, 75, 101499.
- [Background] Lopez, S.M., Martin, F.N., & Thibodeau, L.M. (1997). Performance of monolingual and bilingual speakers of English and Spanish on the Synthetic Sentence Identification Test. American Journal of Audiology, 6(3), 33-38.
- [Background] Fuente A, McPherson B. Auditory processing tests for Spanish-speaking adults: an initial study. Int J Audiol. 2006 Nov;45(11):645-59. doi: 10.1080/14992020600937238. PMID 17118907

RESULTS

PARTICIPANT FLOW:
Pre-assignment Details: Of the 29 enrolled participants, 25 met the inclusion criteria and completed the auditory processing assessments.
Groups:
- L1 First: All participants will receive both interventions (i.e., test materials in English, test materials in Spanish) in a counterbalanced order. Individuals in this arm receive Spanish materials first, then English test materials. Both L1 and L2 assessments will be completed in the same session lasting approximately 3 hours.
- L2 First: All participants will receive both interventions (i.e., test materials in English, test materials in Spanish) in a counterbalanced order. Individuals in this arm receive English materials first, then Spanish test materials. Both L1 and L2 assessments will be completed in the same session lasting approximately 3 hours.
Period: Overall Study
Arm/Group | L1 First | L2 First
Started | 12 | 13
Completed | 12 | 13
Not Completed | 0 | 0

BASELINE CHARACTERISTICS:
Groups:
- Auditory Processing Disorder (APD) Assessment: All participants received both experimental conditions (i.e., test materials in English, test materials in Spanish) in a counterbalanced order.
  English APD assessment: Materials presented in English
  Spanish APD assessment: Materials presented in Spanish
Arm/Group | Auditory Processing Disorder (APD) Assessment
Number analyzed (Participants) | 25
Age, Continuous [Mean (Standard Deviation); unit: years] | 33.48 (11.17)
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 16
  Male | 9
Ethnicity (NIH/OMB) [Count of Participants; unit: Participants]
  Hispanic or Latino | 25
  Not Hispanic or Latino | 0
  Unknown or Not Reported | 0
Race (NIH/OMB) [Count of Participants; unit: Participants]
  American Indian or Alaska Native | 1
  Asian | 0
  Native Hawaiian or Other Pacific Islander | 0
  Black or African American | 0
  White | 11
  More than one race | 4
  Unknown or Not Reported | 9

OUTCOME MEASURES:

1. Primary Outcome: Mean Difference in Scores for APD Assessment Using English vs. Spanish Materials
Description: The APD assessment will include sub-tests (dichotic digits, dichotic word listening test, synthetic sentence identification test). Participants' performance will be scored as percent correct for each sub-test.
Time Frame: 90 minutes
Measure: Mean (Standard Error); unit: percentage of correctly identified stim
Groups:
- APD Assessments: All participants will receive both interventions (i.e., test materials in English, test materials in Spanish) in a counterbalanced order. For analysis, data was pooled across arms since arm assignment was used to mitigate fatigue and/or familiarity effects.
Arm/Group | APD Assessments
Number analyzed (Participants) | 25
percentage of correctly identified stim
  Dichotic Digits - Spanish | 97.40 (0.58)
  Dichotic Digits - English | 94.87 (0.58)
  Dichotic Words - Spanish | 97.14 (0.90)
  Dichotic Words - English | 85.48 (0.90)
  Synthetic Sentences - Spanish | 100 (0)
  Synthetic Sentences - English | 100 (0)
Statistical Analysis 1: Comparison: APD Assessments; Dichotic digits comparison; Test type: Equivalence — The purpose of this study was to evaluate whether the mean performance on auditory processing assessments differed depending on whether the tests were administered in Spanish or English; p < 0.01, Mixed Models Analysis; Slope = -3.89
Statistical Analysis 2: Comparison: APD Assessments; Dichotic words comparison; Test type: Equivalence — [test comment as in outcome 1, analysis 1]; p = 0.69, Mixed Models Analysis; Slope = 5.18

ADVERSE EVENTS:
Time Frame: Participants were monitored for adverse effects during their single study visit which lasted no longer than 3 hours.
Description: No drug or new device was tested during this study. Risk to participants was no greater than what would be experienced in daily life. Established clinical procedures were used and only the language the test was administered in varied.
Arm/Group | Auditory Processing Disorder (APD) Assessment
All-Cause Mortality (participants affected / at risk) | 0/25
Serious Adverse Events (participants affected / at risk) | 0/25
Other Adverse Events (participants affected / at risk) | 0/25

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: No

DOCUMENTS (1):
  • Study Protocol and Statistical Analysis Plan (2023-10-23): https://cdn.clinicaltrials.gov/large-docs/86/NCT05452486/Prot_SAP_000.pdf